CLINICAL TRIAL: NCT00819377
Title: 2- Inhaled Milrinone Prevents the Increase in Pulmonary Artery Pressure After CPB
Brief Title: Milrinone Inhaled in Cardiac Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Andre Denault (Other)
Collaborators: Heart and stoke fondation of Quebec (Unknown); Organon (Industry); Canadian Anesthesiologists' Society (Other)
Responsible Party: Sponsor-Investigator, Andre Denault, MD FRCPC ABIM-CCM, Montreal Heart Institute
Organization: Montreal Heart Institute (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 08-1004
Record Dates: First submitted 2009-01-08; First posted 2009-01-09 (Estimated); Last update posted 2013-10-25 (Estimated); Status verified 2013-10

CONDITIONS: Valvular Stenosis; Valvular Insufficiency; Hypertension, Pulmonary; Coronary Artery Disease
Keywords: Valvular surgery; pulmonary artery pressure
MeSH Terms: conditions — Hypertension, Pulmonary; Coronary Artery Disease | interventions — Milrinone; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Normal saline (Placebo Comparator): Normal saline by inhalation over 15 min
  Interventions: Drug: Normal saline
- Milrinone (Active Comparator): Inhaled milrinone 5 mg(as for the injectable solution)
  Interventions: Drug: Milrinone

INTERVENTIONS:
Drug: Milrinone — inhaled milrinone 5 mg (as for the injectable solution)
  Other Names: Milrinone Cardiac Surgery; Milrinone inhaled; Inhaled milrinone reduces pulmonary artery pressure
  Arms: Milrinone
Drug: Normal saline — 5 ml normal saline by inhalation over 15 min
  Other Names: Placebo; Comparator
  Arms: Normal saline

SUMMARY:
Pulmonary hypertension is an important morbidity factor in patients having to undergo cardiac surgery with cardiopulmonary bypass (ECC). Milrinone used in inhalation, shows evidence of being a pulmonary vasodilator able to possibly contribute to the reduction of pressure on the pulmonary artery.

DETAILED DESCRIPTION:
This controlled, randomized, double-blind study will aim at confirming the efficiency as well as the security of Milrinone, used in inhalation, to diminish the degree of pulmonary hypertension before the cardiopulmonary bypass (ECC) circulation. In addition, the pharmacokinetic and echo graphic repercussions of administering the medication will be analysed. At the present time, there is no data on the pharmacokinetics of the medication when it's administered through inhalation. For this reason, we would like to study the serous rate of the medication in the minutes following its administration through inhalation.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients scheduled for elective valvular or complex (2 or more valves or
* valve and revascularization) cardiac surgery under CPB with preoperative PHT defined as mean pulmonary artery pressure (MPAP) over 30 mmHg or
* systolic pulmonary artery pressure (SPAP) over 40 mmHg (using preoperative right-sided catheterization or estimated by echocardiography).

Exclusion Criteria:

* Cardiac surgery not requiring CPB, contraindication to TEE (esophageal pathology or unstable cervical spine) and emergency surgery.
* Patients will be recruited the day before surgery and randomized using computerized cards by the pharmacy department

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Estimated)
Dates: Start 2009-02; Primary Completion 2012-01 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
To demonstrate that inhaled milrinone administered before CPB is superior to placebo in reducing the severity of difficult separation from bypass | End of CPB

SECONDARY OUTCOMES:
Reduction in morbidity and mortality post-op | At discharge, 3 months, 6 months and 1 year by telephone
Reduction in pulmonary artery pressure | Same day before and after CPB
Right ventricular function measured using transthoracic echocardiography (TTE) and TEE | Same day before and after the CPB
Serum levels of milrinone in relation with the pharmacodynamic marker | Same day pre CPB per CPB and post CPB
reduction of the composite index of hemodynamic complications (defined as hospital death, vasoactive drugs > 24 hours and post-op cardiac arrest), | 24 hrs post op and hospital discharge

CONTACTS AND LOCATIONS:
Overall Officials: Denault André, MD FRCPC, Principal Investigator — Montreal Heart Institute
Locations (1):
- Montreal Heart Institute, Montreal, Quebec, Canada

REFERENCES:
- [Background] Baim DS, McDowell AV, Cherniles J, Monrad ES, Parker JA, Edelson J, Braunwald E, Grossman W. Evaluation of a new bipyridine inotropic agent--milrinone--in patients with severe congestive heart failure. N Engl J Med. 1983 Sep 29;309(13):748-56. doi: 10.1056/NEJM198309293091302. PMID 6888453
- [Background] Denault AY, Lamarche Y, Couture P, Haddad F, Lambert J, Tardif JC, Perrault LP. Inhaled milrinone: a new alternative in cardiac surgery? Semin Cardiothorac Vasc Anesth. 2006 Dec;10(4):346-60. doi: 10.1177/1089253206294400. PMID 17200091
- [Background] Omae T, Kakihana Y, Mastunaga A, Tsuneyoshi I, Kawasaki K, Kanmura Y, Sakata R. Hemodynamic changes during off-pump coronary artery bypass anastomosis in patients with coexisting mitral regurgitation: improvement with milrinone. Anesth Analg. 2005 Jul;101(1):2-8, table of contents. doi: 10.1213/01.ANE.0000155262.37491.6A. PMID 15976197
- [Background] Kikura M, Levy JH, Michelsen LG, Shanewise JS, Bailey JM, Sadel SM, Szlam F. The effect of milrinone on hemodynamics and left ventricular function after emergence from cardiopulmonary bypass. Anesth Analg. 1997 Jul;85(1):16-22. doi: 10.1097/00000539-199707000-00004. PMID 9212116
- [Background] Lobato EB, Florete O Jr, Bingham HL. A single dose of milrinone facilitates separation from cardiopulmonary bypass in patients with pre-existing left ventricular dysfunction. Br J Anaesth. 1998 Nov;81(5):782-4. doi: 10.1093/bja/81.5.782. PMID 10193294
- [Background] Iwagaki T, Irie J, Ijichi K, Uratsuji Y. [The effects of milrinone on hemodynamics in patients undergoing cardiac surgery]. Masui. 2001 Apr;50(4):360-4. Japanese. PMID 11345746
- [Background] Shibata T, Suehiro S, Sasaki Y, Hosono M, Nishi S, Kinoshita H. Slow induction of milrinone after coronary artery bypass grafting. Ann Thorac Cardiovasc Surg. 2001 Feb;7(1):23-7. PMID 11343562
- [Background] Kim JH, Ham BM, Kim YL, Bahk JH, Ryu HG, Jeon YS, Kim KB. Prophylactic milrinone during OPCAB of posterior vessels: implication in angina patients taking beta-blockers. Eur J Cardiothorac Surg. 2003 Nov;24(5):770-6. doi: 10.1016/s1010-7940(03)00393-2. PMID 14583311
- [Background] Hoffman TM, Wernovsky G, Atz AM, Kulik TJ, Nelson DP, Chang AC, Bailey JM, Akbary A, Kocsis JF, Kaczmarek R, Spray TL, Wessel DL. Efficacy and safety of milrinone in preventing low cardiac output syndrome in infants and children after corrective surgery for congenital heart disease. Circulation. 2003 Feb 25;107(7):996-1002. doi: 10.1161/01.cir.0000051365.81920.28. PMID 12600913
- [Background] Maslow AD, Regan MM, Schwartz C, Bert A, Singh A. Inotropes improve right heart function in patients undergoing aortic valve replacement for aortic stenosis. Anesth Analg. 2004 Apr;98(4):891-902. doi: 10.1213/01.ANE.0000107940.23783.33. PMID 15041568
- [Background] Doolan LA, Jones EF, Kalman J, Buxton BF, Tonkin AM. A placebo-controlled trial verifying the efficacy of milrinone in weaning high-risk patients from cardiopulmonary bypass. J Cardiothorac Vasc Anesth. 1997 Feb;11(1):37-41. doi: 10.1016/s1053-0770(97)90250-0. PMID 9058218
- [Background] Yamada T, Takeda J, Katori N, Tsuzaki K, Ochiai R. Hemodynamic effects of milrinone during weaning from cardiopulmonary bypass: comparison of patients with a low and high prebypass cardiac index. J Cardiothorac Vasc Anesth. 2000 Aug;14(4):367-73. doi: 10.1053/jcan.2000.7920. PMID 10972598
- [Background] Solina A, Papp D, Ginsberg S, Krause T, Grubb W, Scholz P, Pena LL, Cody R. A comparison of inhaled nitric oxide and milrinone for the treatment of pulmonary hypertension in adult cardiac surgery patients. J Cardiothorac Vasc Anesth. 2000 Feb;14(1):12-7. doi: 10.1016/s1053-0770(00)90048-x. PMID 10698385
- [Background] Denault AY, Chaput M, Couture P, Hebert Y, Haddad F, Tardif JC. Dynamic right ventricular outflow tract obstruction in cardiac surgery. J Thorac Cardiovasc Surg. 2006 Jul;132(1):43-9. doi: 10.1016/j.jtcvs.2006.03.014. PMID 16798301
- [Background] Couture P, Denault AY, Pellerin M, Tardif JC. Milrinone enhances systolic, but not diastolic function during coronary artery bypass grafting surgery. Can J Anaesth. 2007 Jul;54(7):509-22. doi: 10.1007/BF03022314. PMID 17602036
- [Background] Packer M, Carver JR, Rodeheffer RJ, Ivanhoe RJ, DiBianco R, Zeldis SM, Hendrix GH, Bommer WJ, Elkayam U, Kukin ML, et al. Effect of oral milrinone on mortality in severe chronic heart failure. The PROMISE Study Research Group. N Engl J Med. 1991 Nov 21;325(21):1468-75. doi: 10.1056/NEJM199111213252103. PMID 1944425
- [Background] Cuffe MS, Califf RM, Adams KF Jr, Benza R, Bourge R, Colucci WS, Massie BM, O'Connor CM, Pina I, Quigg R, Silver MA, Gheorghiade M; Outcomes of a Prospective Trial of Intravenous Milrinone for Exacerbations of Chronic Heart Failure (OPTIME-CHF) Investigators. Short-term intravenous milrinone for acute exacerbation of chronic heart failure: a randomized controlled trial. JAMA. 2002 Mar 27;287(12):1541-7. doi: 10.1001/jama.287.12.1541. PMID 11911756
- [Background] Lamarche Y, Malo O, Thorin E, Denault A, Carrier M, Roy J, Perrault LP. Inhaled but not intravenous milrinone prevents pulmonary endothelial dysfunction after cardiopulmonary bypass. J Thorac Cardiovasc Surg. 2005 Jul;130(1):83-92. doi: 10.1016/j.jtcvs.2004.09.011. PMID 15999045
- [Background] Haraldsson s A, Kieler-Jensen N, Ricksten SE. The additive pulmonary vasodilatory effects of inhaled prostacyclin and inhaled milrinone in postcardiac surgical patients with pulmonary hypertension. Anesth Analg. 2001 Dec;93(6):1439-45, table of contents. doi: 10.1097/00000539-200112000-00018. PMID 11726420
- [Background] Sablotzki A, Starzmann W, Scheubel R, Grond S, Czeslick EG. Selective pulmonary vasodilation with inhaled aerosolized milrinone in heart transplant candidates. Can J Anaesth. 2005 Dec;52(10):1076-82. doi: 10.1007/BF03021608. PMID 16326679
- [Background] Bernstein AD, Parsonnet V. Bedside estimation of risk as an aid for decision-making in cardiac surgery. Ann Thorac Surg. 2000 Mar;69(3):823-8. doi: 10.1016/s0003-4975(99)01424-1. PMID 10750767
- [Background] Lamarche Y, Perrault LP, Maltais S, Tetreault K, Lambert J, Denault AY. Preliminary experience with inhaled milrinone in cardiac surgery. Eur J Cardiothorac Surg. 2007 Jun;31(6):1081-7. doi: 10.1016/j.ejcts.2007.02.019. Epub 2007 Apr 2. PMID 17400468
- [Background] Robitaille A, Denault AY, Couture P, Belisle S, Fortier A, Guertin MC, Carrier M, Martineau R. Importance of relative pulmonary hypertension in cardiac surgery: the mean systemic-to-pulmonary artery pressure ratio. J Cardiothorac Vasc Anesth. 2006 Jun;20(3):331-9. doi: 10.1053/j.jvca.2005.11.018. Epub 2006 Apr 19. PMID 16750732
- [Background] Lindsay CA, Barton P, Lawless S, Kitchen L, Zorka A, Garcia J, Kouatli A, Giroir B. Pharmacokinetics and pharmacodynamics of milrinone lactate in pediatric patients with septic shock. J Pediatr. 1998 Feb;132(2):329-34. doi: 10.1016/s0022-3476(98)70454-8. PMID 9506650
- [Background] Oddie CJ, Jackman GP, Bobik A. Analysis of milrinone in plasma using solid-phase extraction and high-performance liquid chromatography. J Chromatogr. 1986 Jan 10;374(1):209-14. doi: 10.1016/s0378-4347(00)83274-0. No abstract available. PMID 3949932
- [Background] Hudson RJ, Thomson IR, Jassal R. Effects of cardiopulmonary bypass on sufentanil pharmacokinetics in patients undergoing coronary artery bypass surgery. Anesthesiology. 2004 Oct;101(4):862-71. doi: 10.1097/00000542-200410000-00010. PMID 15448518
- [Background] Fiset P, Mathers L, Engstrom R, Fitzgerald D, Brand SC, Hsu F, Shafer SL. Pharmacokinetics of computer-controlled alfentanil administration in children undergoing cardiac surgery. Anesthesiology. 1995 Nov;83(5):944-55. doi: 10.1097/00000542-199511000-00006. PMID 7486179
- [Derived] Denault AY, Bussieres JS, Arellano R, Finegan B, Gavra P, Haddad F, Nguyen AQN, Varin F, Fortier A, Levesque S, Shi Y, Elmi-Sarabi M, Tardif JC, Perrault LP, Lambert J. A multicentre randomized-controlled trial of inhaled milrinone in high-risk cardiac surgical patients. Can J Anaesth. 2016 Oct;63(10):1140-1153. doi: 10.1007/s12630-016-0709-8. Epub 2016 Jul 28. PMID 27470232